CLINICAL TRIAL: NCT05737823
Title: Randomised Controlled Feasibility Study and Exploratory Trial of the Carers-ID Intervention: Supporting Family Carers' Mental Health Following the COVID-19 Pandemic
Brief Title: Supporting Family Carers' Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: Baily Thomas Charitable Fund (Unknown); University of Glasgow (Other); University of Sheffield (Other); University of South Wales (Other)
Responsible Party: Principal Investigator, Dr Mark Linden, Reader, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHLS 23_04
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Feasibility
Keywords: Family carer; Intellectual disabilities; Feasibility; Mental health; Intervention
MeSH Terms: conditions — Intellectual Disability; Psychological Well-Being

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Random allocation to the intervention and control conditions will be undertaken by an independent third party not involved with the research. Members of the research team will be blind to allocation to reduce selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carers-ID online support programme (Experimental): Participants in this arm will receive access to the Carers-ID online programme. Participants will be able to access the online programme for 2 weeks.
  Interventions: Behavioral: Carers-ID online support programme
- Wait-list Control (Other): Wait-list control arm
  Interventions: Behavioral: Carers-ID online support programme - Wait-list control

INTERVENTIONS:
Behavioral: Carers-ID online support programme — The Carers-ID online programme, which consists of ten modules which cover topics including: promoting resilience, reducing anxiety, managing stress, accessing local supports, managing family conflict and information for siblings who are carers.
  Arms: Carers-ID online support programme
Behavioral: Carers-ID online support programme - Wait-list control — The same programme as above delivered to the wait-list control after the T2 follow-up data has been collected.
  Arms: Wait-list Control

SUMMARY:
Brief Summary:

Background: Feasibility and acceptability of the Carers-ID intervention to improve mental health outcomes in family carers of people with intellectual disabilities.

Objective:

1. To conduct a Phase II feasibility randomised controlled trial and process evaluation of the Carers-ID programme.
2. To determine the acceptability of outcome measures of stress, anxiety, depression, resilience and well-being in assessing the impact of the programme on family carers.
3. To determine the recruitment and retention rates of participants in the trial.
4. To identify potential effect sizes and estimate appropriate sample size for use in an effectiveness trial.
5. To determine if progression to a phase III effectiveness trial is warranted.

Methodology:

Family carers (n = 120) will be randomised to receive the programme (n=60) or assigned to a wait-list control (n=60) group. The intervention (Carers-ID) consists of ten modules which cover topics including: promoting resilience, reducing anxiety, managing stress, accessing local supports, managing family conflict and information for siblings who are carers. Participants (n=12) who have taken part in the intervention arm of the research will be invited to participate in the process evaluation.

Outcome:

1. Retention of Subjects in Study Assessments (>80% of family carers)
2. Recruitment of Subjects into Study (>90 carers)
3. Acceptability and feasibility of the outcome measures (>80% of family carers)
4. Depression, Anxiety and Stress Scale - 21; The Warwick-Edinburgh Mental Well-being Scale; The Resilience Scale; and The Social Connectedness Scale Revised.

Number of participants to be enrolled: 120 family carers

Main inclusion criteria: Participants will be UK adults >18 years of age and will be caring for a family member with an intellectual disability.

Statistical Analysis: Descriptive statistics will be used to summarise baseline data including demographic variables and questionnaire responses. Inferential statistics (t-tests or ANOVA) will be used as indicators of difference between the intervention and control arms and will be used to determine effect sizes for sample size calculation in a future phase III trial.

Study duration: 24 months

ELIGIBILITY:
Inclusion Criteria:

* Resident of the UK;
* >18 years of age;
* Caring for a family member with an intellectual disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Retention of Subjects in Study Assessments | 3 months
  Retain 80% of intervention and control participants
Recruitment of Subjects Into Study | 3 months
  Sufficient recruitment is set as >90 family carers.
Acceptability and feasibility of the outcome measures | 6 months
  Acceptability and feasibility of the outcome measures determined by process evaluation (>80% of family carers).

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale - 21 (DASS-21) | Baseline (T0), 2 weeks (T1), 3 months (T2)
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, with 21 items in total. Items are rated on a 4 point Likert scale, from 'Did not apply to me at all' to 'Applied to me very much or most of the time'.
  Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items and multiplying by 2, with potential scores ranging from 0 to a maximum of 42. With higher scores indicating increased severity of emotional state.
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Baseline (T0), 2 weeks (T1), 3 months (T2)
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) was developed to enable the measurement of mental wellbeing. The WEMWBS is a 14-item scale of positively worded statements covering feeling and functioning aspects of mental wellbeing. The 14-statements have five response categories from 'none of the time' to 'all of the time'.
  The WEMWBS is scored by summing the scores for each of the 14 items, which are scored from 1 to 5. Scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
The Resilience Scale (RS-25) | Baseline (T0), 2 weeks (T1), 3 months (T2)
  The 25 Item Resilience Scale was developed as a general measure of resilience for adults across the lifespan.
  Participants respond by either agreeing or disagreeing with the statements on a scale of 1(disagree) to 7 (agree). The responses are summed (min 25 to max 175) and a higher score reflects stronger resilience.
The Social Connectedness Scale Revised | Baseline (T0), 2 weeks (T1), 3 months (T2)
  This 20-item scale is used to assess the extent to which persons feel connected to others in their surrounding social area. It is on a Likert scale with 1 being strongly disagree to 6 being strongly agree.
  The negatively worded items are reverse scored and summed together with the positively worded items to create a scale score with a possible range from 20 to 120. An item mean score with a possible range from 1 to 6 can also be calculated by dividing the total scale score by 20 (or the number of scale items). Higher scores on the SCS-R reflect a stronger sense of social connectedness.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University Belfast, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be made available in publications and open access databases.

REFERENCES:
- [Derived] Linden MA, Leonard R, Forbes T, Brown M, Marsh L, Todd S, Hughes N, Truesdale M. Randomised controlled feasibility study protocol of the Carers-ID online intervention to support the mental health of family carers of people with intellectual disabilities. Pilot Feasibility Stud. 2024 Feb 6;10(1):25. doi: 10.1186/s40814-024-01448-w. PMID 38321576
- See also: Carers-ID webpage — https://carers-id.com/